CLINICAL TRIAL: NCT05742399
Title: Clinical Evaluation of the Efficacy and Safety of Novel Drug-free Hyaluronic Acid Topical Nano-carrier in Periocular Rejuvenation
Brief Title: Periocular Rejuvenation by Topical Hyaluronic Acid Nano Particles
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Shimaa Ismail Abdelhamid, Associate professor (MD), Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305360; 00012098 (Other: IRB)
Record Dates: First submitted 2023-01-15; First posted 2023-02-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Tear Trough Eyelid Deformity; Dark Eyelids; Wrinkle
Keywords: periocular; rejuvenation; tear trough; hyaluronic acid; topical; dark circles; wrinkles
MeSH Terms: conditions — Hyperpigmentation of Eyelids

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic acid nanoparticles (2%) (Active Comparator): patients with tear trough will receive hyaluronic acid nano-gel (2%) 2 applications / day (morning and evening) on tear troughs for 1 month
  Interventions: Drug: Hyaluronic acid NanoGel
- Placebo (Placebo Comparator): patients with tear trough will receive placebo conventional gel having the same color, form and packaging for 1 month
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Hyaluronic acid NanoGel — Hyaluronic acid nanoparticles (2%)
  Arms: Hyaluronic acid nanoparticles (2%)
Drug: Placebo gel — conventional gel having the same color, form and packaging
  Arms: Placebo

SUMMARY:
In this study, The investigators aims to evaluate the efficacy and safety of topical hyaluronic acid nanoparticles as a novel nanodermatological tool in periocular rejuvenation as a replacement approach of invasive dermal filler injections.

DETAILED DESCRIPTION:
Tear trough deformity is a main concern of many people (males or females) with age range of 21 to 65 years old or older. Such condition is characterized by a sunken appearance of the eye that results in an aged and dissipated appearance to the eye.Treatment modalities range from camouflage make up, laser resurfacing, platelet-rich plasma therapy, carboxy therapy, mesotherapy, volume augmentation with injectable hyaluronic acid fillers and fat, as well as surgical procedures such as blepharoplasty. Consequently, safe, effective and less invasive treatment options of the tear trough have remained a challenge.

The study will include 30 adult patients (male or female) suffering tear trough deformity.

They will be selected from Dermatology Outpatient Clinic of Alexandria Main University Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 21 and 65 years old
2. Is voluntarily willing to consent to participate in the study
3. Is willing to comply with all requirements of the study including being photographed, follow post treatment care instructions, to attend all treatment, and follow up visits
4. Willingness to waive rights to use of still photos of themselves for research, marketing, or promotional reasons, including on the internet and on social media outlets.
5. Willingness to refrain from other surgical, laser, or injectable treatments in the periorbital region during the entire duration of the study.
6. Ability to provide informed consent.

Exclusion Criteria:

-

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
The efficacy of topical hyaluronic acid nanoparticles in treatment of tear trough | 1 month
  To evaluate the efficacy of topical hyaluronic acid nanoparticles in in treatment of tear trough using Sadick et al scale at baseline and after one month treatment. the score will range from 1-14, in which the higher the score, the worse the outcome
Assessment of improvement of tear trough by topical hyaluronic acid nanoparticles | up to 4 weeks
  Physician assessment will be done at the one-month follow up visit through blinded evaluator-assessed Global Aesthetic Improvement Score. the score will range from 1-5, in which score 1 is associated with best results and score 5 with worst results.
Patient satisfaction of topical hyaluronic acid nanoparticles in treatment of tear trough | 1 month
  Patient satisfaction will be assessed using a visual analogue scale which is ranged from 0-3, 0 is associated with least satisfaction and 3 with the best satisfaction.
Incidence of side effects of topical hyaluronic acid nanoparticles around eyes | up to 4 weeks
  Incidence of side effects will be evaluated at all visits by reporting any adverse events such as erythema, dryness, itching, edema or hyperpigmentation.

SECONDARY OUTCOMES:
The efficacy of topical hyaluronic acid nanoparticles in treatment of dark circles | up to 4 weeks
  To evaluate the efficacy of topical hyaluronic acid nanoparticles in treatment of of dark circles according to the intenisty of pigmentaion (mild, moderate or intense)

OTHER OUTCOMES:
The efficacy of topical hyaluronic acid nanoparticles in treatment of periocular wrinkles | 1 month
  To evaluate the efficacy of topical hyaluronic acid nanoparticles in treatment of wrinkles according to Glogau wrinkles scale at baseline and after one month treatment. it ranges from 1-4. one mean youngest and 4 means oldest

CONTACTS AND LOCATIONS:
Overall Officials: Yosra S.R Elnaggar, MD, Study Chair — Alexandria University
Locations (1):
- Shaimaa Ismail Omar, Alexandria, Elazarita, Egypt

IPD SHARING:
Plan to Share IPD: No
Because we will publish the study in a journal

REFERENCES:
- [Background] 1. Diab HM, Elhosseiny R, Bedair NI, Khorkhed AH. Efficacy and safety of plasma gel versus platelet-rich plasma in periorbital rejuvenation: a comparative split-face clinical and Antera 3D camera study. Archives of dermatological research. 2021. 2. Sharad J. Dermal Fillers for the Treatment of Tear Trough Deformity: A Review of Anatomy, Treatment Techniques, and their Outcomes. Journal of cutaneous and aesthetic surgery. 2012;5(4):229-38. 3. Viana GA, Osaki MH, Cariello AJ, Damasceno RW, Osaki TH. Treatment of the tear trough deformity with hyaluronic acid. Aesthetic surgery journal. 2011;31(2):225-31. 4. Hirmand H. Anatomy and nonsurgical correction of the tear trough deformity. Plastic and reconstructive surgery. 2010;125(2):699-708. 5. Shah-Desai S, Joganathan V. Novel technique of non-surgical rejuvenation of infraorbital dark circles. Journal of cosmetic dermatology. 2021;20(4):1214-20. 6. Trinh LN, Grond SE, Gupta A. Dermal Fillers for Tear Trough Rejuvenation: A Systematic Review. Facial plastic surgery : FPS. 2021. 7. Lubart R, Yariv I, Fixler D, Lipovsky A. Topical Hyaluronic Acid Facial Cream with New Micronized Molecule Technology Effectively Penetrates and Improves Facial Skin Quality: Results from In-vitro, Ex-vivo, and In-vivo (Open-label) Studies. The Journal of clinical and aesthetic dermatology. 2019;12(10):39-44. 8. Chiari-Andréo BG, Almeida-Cincotto MGJd, Oshiro JA, Taniguchi CYY, Chiavacci LA, Isaac VLB. Chapter 5 - Nanoparticles for cosmetic use and its application. In: Grumezescu AM, editor. Nanoparticles in Pharmacotherapy: William Andrew Publishing; 2019.113-46.